CLINICAL TRIAL: NCT01838590
Title: A Phase 3, Randomized, Open-Label, Study to Evaluate the Safety and Efficacy of Sofosbuvir Plus Ribavirin Administered for Either 12 or 24 Weeks in Treatment-Naïve and Treatment-Experienced Egyptian Adults With Chronic Genotype 4 HCV Infection.
Brief Title: Sofosbuvir Plus Ribavirin Administered for Either 12 or 24 Weeks in Treatment-Naive and Treatment-Experienced Egyptian Adults With Chronic Genotype 4 Hepatitis C Virus (HCV) Infection
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-334-0138
Record Dates: First submitted 2013-04-15; First posted 2013-04-24 (Estimated); Results first posted 2015-05-22 (Estimated); Last update posted 2015-05-22 (Estimated); Status verified 2015-05

CONDITIONS: Hepatitis C Virus
Keywords: Liver Diseases; Digestive System Diseases; Hepatitis, Viral, Human; Virus Diseases; Enterovirus Infections; Picornaviridae Infections; RNA Virus Infections; Flaviviridae Infections; Antiviral Agents; Anti-Infective Agents; Therapeutic Uses; Pharmacologic Actions; Antimetabolites; Molecular Mechanisms of Pharmacological Action; HCV genotype 4 (GT-4); HCV; Sustained Virologic Response; Direct Acting Antiviral; Combination Therapy; GS-7977; Ribavirin; Open Label; Sofosbuvir; Additional relevant MeSH terms:; Hepatitis; Hepatitis, Chronic; Hepatitis C; Hepatitis C, Chronic
MeSH Terms: conditions — Hepatitis C; Liver Diseases; Digestive System Diseases; Hepatitis, Viral, Human; Virus Diseases; Enterovirus Infections; Picornaviridae Infections; RNA Virus Infections; Flaviviridae Infections; Hepatitis; Hepatitis, Chronic; Hepatitis C, Chronic | interventions — Sofosbuvir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- SOF+RBV 12 Weeks (Experimental): Participants will receive SOF+RBV for 12 weeks.
  Interventions: Drug: SOF; Drug: RBV
- SOF+RBV 24 Weeks (Experimental): Participants will receive SOF+RBV for 24 weeks.
  Interventions: Drug: SOF; Drug: RBV

INTERVENTIONS:
Drug: SOF — Sofosbuvir (SOF) 400 mg tablet administered orally once daily
  Other Names: Sovaldi®; GS-7977
Drug: RBV — Ribavirin (RBV) 200 mg tablets administered orally in a divided daily dose (< 75 kg = 1000 mg and ≥ 75 kg = 1200 mg)

SUMMARY:
This study is to to evaluate the safety, tolerability, and efficacy of sofosbuvir (SOF) plus ribavirin (RBV) in Egyptian adults with genotype 4 hepatitis C virus (HCV) infection.

ELIGIBILITY:
Inclusion Criteria:

* Treatment experienced and naïve subjects
* Chronic genotype 4 HCV-infection
* Not co-infected with HIV
* Screening laboratory values within defined thresholds
* Use of highly effective contraception methods
* Subject must be able to comply with the dosing instructions for study drug administration and able to complete the study schedule of assessments.

Exclusion Criteria:

* History of any other clinically significant chronic liver disease
* Pregnant or nursing female or male with pregnant female partner
* History of clinically-significant illness or any other major medical disorder that may interfere with subject treatment, assessment or compliance with the protocol
* Excessive alcohol ingestion or significant drug abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2013-03; Primary Completion 2014-05 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn Kersey, Study Director — Gilead Sciences
Locations (2):
- Egypt (2):
  - Al Mansurah
  - Cairo

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at a total of 3 study sites in Egypt. The first participant was screened on 30 March 2013. The last study visit occurred on 04 August 2014.
Pre-assignment Details: 141 participants were screened.
Groups:
- SOF+RBV 12 Weeks: Sofosbuvir (SOF) 400 mg tablet once daily + ribavirin (RBV) tablets (1000-1200 mg daily based on weight) for 12 weeks
- SOF+RBV 24 Weeks: SOF 400 mg tablet once daily + RBV tablets (1000-1200 mg daily based on weight) for 24 weeks
Period: Overall Study
Arm/Group | SOF+RBV 12 Weeks | SOF+RBV 24 Weeks
Started | 52 | 51
Completed | 40 | 46
Not Completed | 12 | 5
Not completed — Lack of Efficacy | 12 | 4
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set: participants who were randomized and received at least 1 dose of study drug
Groups:
- SOF+RBV 12 Weeks, TN: SOF 400 mg tablet once daily + RBV tablets (1000-1200 mg daily based on weight) for 12 weeks (treatment naive (TN))
- SOF+RBV 12 Weeks, TE: SOF 400 mg tablet once daily + RBV tablets (1000-1200 mg daily based on weight) for 12 weeks (treatment experienced (TE))
- SOF+RBV 24 Weeks, TN: SOF 400 mg tablet once daily + RBV tablets (1000-1200 mg daily based on weight) for 24 weeks (treatment naive)
- SOF+RBV 24 Weeks, TE: SOF 400 mg tablet once daily + RBV tablets (1000-1200 mg daily based on weight) for 24 weeks (treatment experienced)
- Total: Total of all reporting groups
Arm/Group | SOF+RBV 12 Weeks, TN | SOF+RBV 12 Weeks, TE | SOF+RBV 24 Weeks, TN | SOF+RBV 24 Weeks, TE | Total
Number analyzed (Participants) | 25 | 27 | 24 | 27 | 103
Age, Continuous [Mean (Standard Deviation); unit: years] | 43 (12.3) | 46 (11.5) | 46 (14.5) | 51 (8.3) | 47 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 8 | 11 | 8 | 34
  Male | 18 | 19 | 13 | 19 | 69
Race/Ethnicity, Customized [Number; unit: participants]
  White | 25 | 27 | 24 | 27 | 103
Race/Ethnicity, Customized [Number; unit: participants]
  Not Hispanic or Latino | 25 | 27 | 24 | 27 | 103
Cirrhosis Status [Number; unit: participants]
  No | 22 | 22 | 21 | 21 | 86
  Yes | 3 | 5 | 3 | 6 | 17
IL28b Status [Number; unit: participants] — CC, CT, and TT alleles are different forms of the IL28b gene.
  participants
    CC | 8 | 1 | 6 | 5 | 20
    CT | 12 | 18 | 12 | 21 | 63
    TT | 5 | 8 | 6 | 1 | 20
HCV RNA [Mean (Standard Deviation); unit: log10 IU/mL] | 5.6 (0.73) | 5.9 (0.57) | 5.5 (0.75) | 6.2 (0.49) | 5.8 (0.70)
HCV RNA Category [Number; unit: participants]
  < 800,000 IU/mL | 15 | 11 | 15 | 8 | 49
  ≥ 800,000 IU/mL | 10 | 16 | 9 | 19 | 54

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Sustained Virologic Response (SVR) at 12 Weeks After Discontinuation of Therapy (SVR12)
Description: SVR12 was defined as HCV RNA < the lower limit of quantitation (LLOQ; ie, 25 IU/mL) at 12 weeks after stopping study treatment.
Time Frame: Posttreatment Week 12
Population: Full Analysis Set: participants with genotype 4 HCV infection who were randomized and received at least one dose of study drug
Measure: Number; unit: percentage of participants
Groups:
- SOF+RBV 12 Weeks, TN: SOF 400 mg tablet once daily + RBV tablets (1000-1200 mg daily based on weight) for 12 weeks (treatment naive)
- SOF+RBV 12 Weeks, TE: SOF 400 mg tablet once daily + RBV tablets (1000-1200 mg daily based on weight) for 12 weeks (treatment experienced)
Arm/Group | SOF+RBV 12 Weeks, TN | SOF+RBV 12 Weeks, TE | SOF+RBV 24 Weeks, TN | SOF+RBV 24 Weeks, TE
Number analyzed (Participants) | 25 | 27 | 24 | 27
percentage of participants | 84.0 | 70.4 | 91.7 | 88.9

2. Primary Outcome: Percentage of Participants Who Permanently Discontinued Any Study Drug Due to an Adverse Event
Time Frame: Up to 24 weeks
Population: Safety Analysis Set: participants who were randomized and received at least 1 dose of study drug
Measure: Number; unit: percentage of participants
Groups:
- SOF+RBV 12 Weeks: SOF 400 mg tablet once daily + RBV tablets (1000-1200 mg daily based on weight) for 12 weeks
Arm/Group | SOF+RBV 12 Weeks | SOF+RBV 24 Weeks
Number analyzed (Participants) | 52 | 51
percentage of participants | 0 | 0

3. Secondary Outcome: Percentage of Participants With Sustained Virologic Response at 4 and 24 Weeks After Discontinuation of Therapy (SVR4 and SVR24)
Description: SVR4 and SVR 24 were defined as HCV RNA < LLOQ at 4 and 24 weeks following the last dose of study drug, respectively.
Time Frame: Posttreatment Weeks 4 and 24
Population: Full Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | SOF+RBV 12 Weeks, TN | SOF+RBV 12 Weeks, TE | SOF+RBV 24 Weeks, TN | SOF+RBV 24 Weeks, TE
Number analyzed (Participants) | 25 | 27 | 24 | 27
percentage of participants
  SVR4 | 88.0 | 74.1 | 91.7 | 88.9
  SVR24 | 84.0 | 70.4 | 91.7 | 88.9

4. Secondary Outcome: Percentage of Participants Experiencing On-treatment Virologic Failure
Description: On-treatment virologic failure was defined as
  * Breakthrough (confirmed HCV RNA ≥ LLOQ after having previously had HCV RNA < LLOQ while on treatment), or
  * Rebound (confirmed > 1 log10 IU/mL increase in HCV RNA from nadir while on treatment), or
  * Non-response (HCV RNA persistently ≥ LLOQ through 8 weeks of treatment)
Time Frame: Up to 24 weeks
Population: Full Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | SOF+RBV 12 Weeks, TN | SOF+RBV 12 Weeks, TE | SOF+RBV 24 Weeks, TN | SOF+RBV 24 Weeks, TE
Number analyzed (Participants) | 25 | 27 | 24 | 27
percentage of participants | 0 | 0 | 0 | 0

5. Secondary Outcome: Percentage of Participants Experiencing Virologic Relapse
Description: Virologic relapse was defined as confirmed HCV RNA ≥ LLOQ during the posttreatment period having achieved HCV RNA < LLOQ at last on-treatment visit.
Time Frame: Up to Posttreatment Week 24
Population: Full Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | SOF+RBV 12 Weeks, TN | SOF+RBV 12 Weeks, TE | SOF+RBV 24 Weeks, TN | SOF+RBV 24 Weeks, TE
Number analyzed (Participants) | 25 | 27 | 24 | 27
percentage of participants | 16.0 | 29.6 | 4.2 | 11.1

ADVERSE EVENTS:
Time Frame: Up to 24 weeks plus 30 days
Description: Safety Analysis Set
Arm/Group | SOF+RBV 12 Weeks | SOF+RBV 24 Weeks
Serious Adverse Events (participants affected / at risk) | 0/52 | 2/51
Other Adverse Events (participants affected / at risk) | 34/52 | 38/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SOF+RBV 12 Weeks (N=52) | SOF+RBV 24 Weeks (N=51)
Cerebral Ischaemia (Nervous system disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | SOF+RBV 12 Weeks (N=52) | SOF+RBV 24 Weeks (N=51)
Anaemia (Blood and lymphatic system disorders) | 6 | 10
Dyspepsia (Gastrointestinal disorders) | 4 | 8
Abdominal pain upper (Gastrointestinal disorders) | 6 | 3
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 | 5
Abdominal pain (Gastrointestinal disorders) | 2 | 3
Diarrhoea (Gastrointestinal disorders) | 1 | 4
Nausea (Gastrointestinal disorders) | 1 | 4
Constipation (Gastrointestinal disorders) | 4 | 0
Vomiting (Gastrointestinal disorders) | 1 | 3
Fatigue (General disorders) | 7 | 14
Pyrexia (General disorders) | 2 | 3
Nasopharyngitis (Infections and infestations) | 1 | 3
Bone pain (Musculoskeletal and connective tissue disorders) | 4 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 3
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 3
Headache (Nervous system disorders) | 6 | 11
Somnolence (Nervous system disorders) | 2 | 3
Insomnia (Psychiatric disorders) | 7 | 10
Renal colic (Renal and urinary disorders) | 0 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 5
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 | 6
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years